CLINICAL TRIAL: NCT04594551
Title: Immunogenicity and Safety of the Purified Vero Rabies Vaccine - Serum Free (VRVg) Using the Zagreb Regimen as Simulated Rabies Post-exposure Prophylaxis in Healthy Adults in Thailand
Brief Title: Study of Purified Vero Rabies Vaccine Compared With a Reference Rabies Vaccine as Simulated Rabies Post-Exposure Prophylaxis in Adults in Thaïland
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VRV00014; U1111-1238-1726 (Other: UTN)
Record Dates: First submitted 2020-10-12; First posted 2020-10-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rabies (Healthy Volunteers)
Keywords: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: VRVg-2 + HRIG (Experimental): VRVg-2 4 injections: 2 at Day 0, 1 at Day 7, 1 at Day 21
  + HRIG at D0
  Interventions: Biological: Purified vero rabies vaccine - serum free; Biological: Human rabies immunoglobulins
- Group 2: Verorab + HRIG (Active Comparator): Verorab 4 injections: 2 at Day 0, 1 at Day 7, 1 at Day 21
  + HRIG at D0
  Interventions: Biological: Purified inactivated rabies vaccine; Biological: Human rabies immunoglobulins

INTERVENTIONS:
Biological: Purified vero rabies vaccine - serum free — Pharmaceutical form:freeze-dried - Route of administration: intramuscular
  Other Names: VRVg-2
  Arms: Group 1: VRVg-2 + HRIG
Biological: Purified inactivated rabies vaccine — Pharmaceutical form:freeze-dried - Route of administration: intramuscular
  Other Names: Verorab
  Arms: Group 2: Verorab + HRIG
Biological: Human rabies immunoglobulins — Pharmaceutical form:liquid/solution in 2 mL vials - Route of administration: intramuscular
  Other Names: HRIG

SUMMARY:
Primary Objective:

To describe the immune response induced by VRVg-2 and Verorab vaccines at D14 and D35 when co-administered with Human Rabies Immunoglobulins (HRIG) at D0, according to the Zagreb (2-1-1) IM regimen in healthy adult subjects.

Secondary Objective:

Immunogenicity To describe the immune response induced by VRVg-2 and Verorab vaccines at D90 when co-administered with HRIG at D0, according to the Zagreb (2-1-1) IM regimen in healthy adult subjects.

Safety To describe the safety profile of VRVg-2 and Verorab vaccines when co administered with HRIG at D0, after each vaccination.

DETAILED DESCRIPTION:
The duration of each subject's participation in the study will be approximately 7 months (21 day-vaccination period followed by 6 months safety follow-up period).

ELIGIBILITY:
Inclusion criteria :

* Aged ≥ 18 years on the day of inclusion
* Able to attend all scheduled visits and to comply with all study procedures
* Body Mass Index (BMI): 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2s

Exclusion criteria:

* Subject is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and 1 month after each vaccination. To be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment or, planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks (28 days) preceding the first study vaccination or planned receipt of any vaccine prior to Visit 7 (D90)
* Previous vaccination against rabies (in pre- or post-exposure regimen) with either the study vaccines or another vaccine
* Bite by, or exposure to a potentially rabid animal in the previous 6 months without post-exposure prophylaxis
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* At high risk for rabies exposure
* Known systemic hypersensitivity to any of the study/control vaccine components or to human rabies immunoglobulin (HRIG), or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Personal history of Guillain-Barré syndrome
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Receipt of chloroquine or hydroxychloroquine up to 2 months prior to the study or through to study until Visit 7

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-10-11 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving rabies virus neutralizing antibody (RVNA) titer greater than or equal to (≥) 0.5 IU/mL | Day 14 (post-vaccination)
  RVNA titers will be measured by rapid fluorescent focus inhibition test (RFFIT)
Percentage of participants achieving RVNA titer greater than or equal to (≥) 0.5 IU/mL | Day 35 (post-vaccination)
  RVNA titers will be measured by RFFIT
Number of Participants achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 14 (post-vaccination)
  RVNA titers will be measured by RFFIT - Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Number of Participants achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 35 (post-vaccination)
  RVNA titers will be measured by RFFIT - Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) | Day 14 (post-vaccination
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 14 - RVNA ratios Day14/Day0 will be calculated
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) | Day 35 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 35 - RVNA ratios Day35/Day0 will be calculated

SECONDARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systematic AEs
Percentage of participants reporting solicited injection site and systemic reactions | Within 7 days post-vaccination
  Solicited injection site reactions:
  - pain, erythema, and swelling in adults (aged ≥ 18 years)
  Solicited systemic reactions:
  - fever, headache, malaise and myalgia in adults (aged ≥ 18 years)
Number of participants reporting unsolicited injection site AEs | Within 28 days post-vaccination
  Unsolicited injection site AEs
Number of participants reporting unsolicited systemic AEs | Between each vaccination and up to 28 days after the last vaccination
  Unsolicited systemic AEs
Number of participants reporting serious adverse events (SAEs) | Up to 6 months after last vaccination
  SAEs, including adverse event of special interest (AESIs)
Percentage of participants achieving rabies virus neutralizing antibody (RVNA) titer greater than or equal to (≥) 0.5 IU/mL | Day 90 (post-vaccination)
  RVNA titers will be measured by RFFIT
Number of Participants achieving RVNA titer greater than or equal to (≥) lower limit of quantification | Day 90 (post-vaccination)
  RVNA titers will be measured by RFFIT - Lower limit of quantification for RFFIT assay is 0.2 IU/mL
Geometric Mean Titer Ratio (GMTR) of individual RVNA titer: (post-/pre-vaccination) | Day 90 (post-vaccination)
  RVNA titers against rabies virus will be measured by RFFIT at Day 0 and Day 90 - RVNA ratios Day90/Day0 will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Thailand (3):
  - Investigational site number 7640002, Bangkok
  - Investigational site number 7640001, Bangkok
  - Investigational site number 7640003, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VRV00014 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25381&tenant=MT_SNY_9011